CLINICAL TRIAL: NCT03566199
Title: An Open Label Single Arm Phase I/II Study of MTX110 Delivered by Convection-enhanced Delivery (CED) in Patients With Diffuse Intrinsic Pontine Glioma (DIPG) Previously Treated With External Beam Radiation Therapy
Brief Title: MTX110 by Convection-Enhanced Delivery in Treating Participants With Newly-Diagnosed Diffuse Intrinsic Pontine Glioma
Acronym: PNOC015
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: Midatech Pharma US Inc. (Industry); Pacific Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Assistant Professor of Clinical Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170817; NCI-2018-01085 (Registry Identifier: Clinical Trials Reporting Program (CTRP)); PNOC015 (Other: Pacific Pediatric Neuro-Oncology Consortium (PNOC))
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (MTX110) (Experimental): Participants receive panobinostat nanoparticle formulation MTX110 IT by CED infusion on day 1 or days 1 and 2 as determined by dose level. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Panobinostat Nanoparticle Formulation MTX110; Drug: Convection-Enhanced Delivery (CED)

INTERVENTIONS:
Drug: Panobinostat Nanoparticle Formulation MTX110 — Given IT
  Other Names: MTX-110; MTX110 (CN)
Drug: Convection-Enhanced Delivery (CED) — Undergo CED
  Other Names: CED

SUMMARY:
This phase I/II trial studies the side effects of panobinostat nanoparticle formulation MTX110 (MTX110) in treating participants with newly-diagnosed diffuse intrinsic pontine glioma. Panobinostat nanoparticle formulation MTX110 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of repeated administration of MTX110 co-infused with gadoteridol given by intratumoral convection enhanced delivery in children with newly diagnosed diffuse intrinsic pontine glioma (DIPG).

SECONDARY OBJECTIVES:

I. To determine the clinical efficacy of repeated administration of MTX110 given by intratumoral convection-enhanced delivery (CED) in children with newly diagnosed DIPG in the confines of a phase I and early efficacy study.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Participants receive panobinostat nanoparticle formulation MTX110 intratumorally (IT) by CED infusion on day 1 or days 1 and 2 as determined by dose level. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment participants are followed up at 30 days and then every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed DIPG by magnetic resonance imaging (MRI); defined as patients with a pontine location and diffuse involvement of at least 2/3 of the pons are eligible without histologic diagnosis. For lesions with typical imaging features, biopsy is neither encouraged nor required for eligibility. Tumors that are biopsied will be eligible if proven to be supportive of the diagnosis of a DIPG. Consensus of diagnosis by the study team must be met.
* Patients who have completed focal radiotherapy within 14 weeks from time of enrollment are eligible.
* Treatment must begin at a minimum of 4 weeks after, but no later than 14 weeks after, the date of completion of focal radiotherapy.
* Prior chemotherapy: Patients should be at least 30 days from last chemotherapy dose prior to start of CED infusion, with exception of antibody half-lives. For antibody therapies, at least 3 half-lives of the antibody after last dose of monoclonal antibody should have passed prior to CED infusion. Patients less than 30 days from last chemotherapy dose should be discussed with the study chair(s).
* Prior radiation: Patients must have received prior treatment with focal radiotherapy as part of initial treatment for DIPG and had their last dose at least 4 weeks prior to and no later than 14 weeks from the first CED treatment. Standard focal radiation therapy will include 54 to 60 Gy by external beam radiotherapy to the brainstem.
* Age ≥ 2 years of age to 21 years. Patients younger than 3 years of age may be enrolled on study at the discretion of the Study Chair(s) if supporting evidence that brainstem lesion represents a brainstem glioma.
* Karnofsky Performance Score ≥ 50 for patients > 16 years of age and Lansky Performance Score ≥ 50 for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are able to mobilize using a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Life expectancy of greater than 12 weeks measured from the date of completion of radiotherapy.
* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm^3.
* Hemoglobin ≥ 8g/dl.
* Platelet count ≥ 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Normal coagulation defined as normal International Normalized Ratio (INR) or per institutional guidelines.
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 milliliters (mL)/minute (min)/1.73 m^2.
* A serum creatinine (mg/dL) based on age/gender as follows:

  * Age: 2 to < 6 years; Male: 0.8; Female: 0.8
  * Age: 6 to < 10 years; Male: 1; Female: 1
  * Age: 10 to < 13 years; Male: 1.2; Female: 1.2
  * Age: 13 to < 16 years; Male:1.5; Female: 1.4
  * Age ≥ 16 years; Male: 1.7; Female: 1.4
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age.
* Serum glutamate pyruvate transaminase (SGPT) [alanine aminotransferase (ALT)] ≤ 110 U/L.
* Serum albumin ≥ 2 g/dL.
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled.
* The effects of MTX110 on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of MTX110 injection administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Able to understand, and willing to sign, a written informed consent document.
* Patients who are unable to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Exclusion Criteria:

* Patients who had clinical and/or radiographic (MRI) progression of tumor following external beam radiation therapy.
* Patients with metastatic disease, including leptomeningeal or subarachnoid disseminated disease.
* Patients with tumor morphology that predicts poor coverage of the majority of the tumor including bilateral thalamic involvement, or cysts that represent > 50% of cross-sectional areas of the pons. These subjects should be discussed with the study chairs.
* Patients who are receiving any other investigational agents or other tumor-directed therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MTX110 or gadolinium.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 14 days of registration.
* Patients with MRI or clinical evidence of uncontrolled tumor mass effect are excluded; the assessment of mass effect should be made by the study chairs and study neurosurgeons prior to any planned CED treatment.
* Untreated symptomatic hydrocephalus determined by treating physician.
* Patients with evidence of intra-tumoral hemorrhage > 5 mm maximal diameter. These subjects should be discussed with the study chair.
* Subjects with prolonged corrected QT (QTc) (> 450 msec) will be excluded from the study.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were only enrolled into Phase 1 of the clinical trial. The phase 2 expansion cohort was not activated for enrollment at behest of pharmaceutical supplier.
Pre-assignment Details: Each participant was permitted to have a dose-escalation assigned to subsequent rounds of CED treatment upon review of safety data at each round. A dose-escalation during treatment in a previous participant, determined the starting dosage assigned to the next participant. The first three participants enrolled received escalated doses in the second or third round of CED treatment.
Groups:
- Phase 1: Starting Dose Level 1 (MTX110): Participant received starting dose of single CED of 30 micrometer of MTX110 on 1 day (day 1); Total volume 3 mL. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 1: Starting Dose Level 2 (MTX110): Participant received starting dose of repeated CED of 30 micrometer of MTX110 on n 2 consecutive days (days 1, 2); Total volume 6 mL (3 mL on each day).
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 1: Starting Dose Level 3 (MTX110): Participant received starting dose of repeated CED of 30 micrometer of MTX110 on n 2 consecutive days (days 1, 2); Total volume 8 mL (4 mL on each day).
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 1: Starting Dose Level 4 (MTX110): Participant received starting dose of repeated CED of 30 micrometer of MTX110 on n 2 consecutive days (days 1, 2); Total volume 10 mL (5 mL on each day).
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 1: Starting Dose Level 5 (MTX110): Participant received starting dose of repeated CED of 30 micrometer of MTX110 on n 2 consecutive days (days 1, 2); Total volume 12 mL (6 mL on each day).
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 1: Starting Dose Level 6 (MTX110): Participant received starting dose of repeated CED of 60 micrometer of MTX110 on n 2 consecutive days (days 1, 2); Total volume 12 mL (6 mL on each day).
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 1: Starting Dose Level 7 (MTX110): Participant received starting dose of repeated CED of 90 micrometer of MTX110 on n 2 consecutive days (days 1, 2); Total volume 12 mL (6 mL on each day).
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
- Phase 2: Participants will receive Recommended Phase 2 Dose (RP2D)
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
Period: Overall Study
Arm/Group | Phase 1: Starting Dose Level 1 (MTX110) | Phase 1: Starting Dose Level 2 (MTX110) | Phase 1: Starting Dose Level 3 (MTX110) | Phase 1: Starting Dose Level 4 (MTX110) | Phase 1: Starting Dose Level 5 (MTX110) | Phase 1: Starting Dose Level 6 (MTX110) | Phase 1: Starting Dose Level 7 (MTX110) | Phase 2
Started | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Completed | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: While individual participants were assigned to receive separate doses, participants are presented in one Arm/Group due to confidentiality concerns for this rare disease study
Groups:
- Phase 1: Treatment (MTX110) - All Participants: Participants receive panobinostat nanoparticle formulation MTX110 IT by CED infusion on day 1 or days 1 and 2 as determined by dose level. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Panobinostat Nanoparticle Formulation MTX110: Given IT Convection-Enhanced Delivery (CED): Undergo CED
Arm/Group | Phase 1: Treatment (MTX110) - All Participants
Number analyzed (Participants) | 7
Age, Customized [Median (Full Range); unit: years] | 8 [5 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Grade 3 or Higher, Treatment-related, Adverse Events
Description: Adverse events and clinically significant laboratory abnormalities which meet Grade 3, 4, or 5 criteria according to Common Terminology Criteria for Adverse Events (CTCAE) classified by investigators and treating physicians as related to study treatment (probable, possible, and definite) will be summarized by maximum intensity/grade. Adverse events will be graded according to CTCAE version 4.0.
Time Frame: Up to 12 Months
Population: as for baseline characteristics
Measure: Number; unit: proportion of participants
Groups:
- Phase 1: Treatment (MTX110): Participants receive panobinostat nanoparticle formulation MTX110 IT by CED infusion on day 1 or days 1 and 2 as determined by dose level. Courses repeat every 4-8 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Panobinostat Nanoparticle Formulation MTX110: Given IT
  Convection-Enhanced Delivery (CED): Undergo CED
Arm/Group | Phase 1: Treatment (MTX110)
Number analyzed (Participants) | 7
proportion of participants
  Muscle weakness right-sided (Grade 3) | 0.142
  Stridor (Grade 3) | 0.142
  Vagus nerve disorder (Grade 3) | 0.142
  Gait disturbance (Grade 3) | 0.142
  Neutrophil count decreased (Grade 3) | 0.142

2. Secondary Outcome: Overall Survival Rate (OS) at 12 Months
Description: Overall survival is defined as the percentage of participants alive from time of diagnosis up to 12 months.
Time Frame: Up to 12 Months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Treatment (MTX110)
Number analyzed (Participants) | 7
percentage of participants | 85.7 [63.3 to 100]

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Additional adverse event and mortality data was collected for participants for up to 24 months following initial diagnosis. While individual participants were assigned to receive separate doses, participants are presented in one Arm/Group due to confidentiality concerns for this rare disease study.
Arm/Group | Phase 1: Treatment (MTX110)
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Treatment (MTX110) (N=7)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Vagus nerve disorder (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Treatment (MTX110) (N=7)
Fatigue (General disorders) | 4 (5)
Gait disturbance (General disorders) | 3 (5)
Pain (General disorders) | 3 (8)
Irritability (General disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (8)
Ataxia (Nervous system disorders) | 4 (17)
Dizziness (Nervous system disorders) | 4 (5)
Abducens nerve disorder (Nervous system disorders) | 3 (4)
Dysarthria (Nervous system disorders) | 2 (7)
Facial nerve disorder (Nervous system disorders) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 2 (4)
Paresthesia (Nervous system disorders) | 2 (2)
Trigeminal nerve disorder (Nervous system disorders) | 2 (2)
Vagus nerve disorder (Nervous system disorders) | 2 (2)
Accessory nerve disorder (Nervous system disorders) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 3 (9)
White blood cell decreased (Investigations) | 3 (8)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (5)
Weight loss (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 4 (7)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Corneal ulcer (Eye disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Phase 2 expansion cohort was not activated at behest of pharmaceutical supplier.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03566199/Prot_SAP_000.pdf